CLINICAL TRIAL: NCT06544044
Title: Efficacy of Brief Mindfulness Based Self-Compassion Intervention for Management of Anger Among Adolescents
Brief Title: Efficacy of Brief Mindfulness Based Self- Compassion Intervention for Management of Anger Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Noor (Other)
Collaborators: Fatima Jinnah Women University (Other)
Responsible Party: Sponsor-Investigator, Fatima Noor, Student, Fatima Jinnah Women University
Organization: Fatima Jinnah Women University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FJWU/EC/2024/81
Record Dates: First submitted 2024-07-20; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Aggression
Keywords: Aggression; Self Compassion; Adolescent
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapist (Experimental): The only one researcher, an experienced mindfulness practitioner and group therapist, leads groups of 10-15 students in weekly 90-minute sessions to deliver the program.
  Interventions: Behavioral: Brief Mindfulness' Self compassion

INTERVENTIONS:
Behavioral: Brief Mindfulness' Self compassion — session includes mindfulness exercises like breath awareness and body scans, self-compassion practices like self-kindness meditations, and emotional regulation strategies such as cognitive reappraisal and response modulation. Discussions focus on applying mindfulness and self-compassion to manage difficult emotions, improve interpersonal interactions, and reduce aggression. Home practice assignments encourage students to integrate mindfulness and self-compassion into their daily lives. The program curriculum is based on existing evidence-based interventions, including mindfulness-based stress reduction for teens.

SUMMARY:
This study investigates the effectiveness of a short self-compassion mental intervention in reducing aggression among adolescents. Although they display potential, current solutions are arduous and time-consuming. The study provides preliminary results on the effectiveness of this method in addressing the lack of information. The intervention's simplicity and precision have the potential to greatly influence the treatment of teenage violence. This could lead to the general acceptance and implementation of mindfulness-based self-compassion, making it accessible at a reasonable cost. The study's brevity and specificity hold promise for broader implementation. A significant gap exists in the literature concerning brief mindfulness-based self-compassion interventions tailored specifically to address adolescent aggression. Most existing studies have explored more extended interventions or general mindfulness programs, leaving a dearth of research on the effectiveness of concise, targeted interventions for adolescents dealing with aggression.

DETAILED DESCRIPTION:
The study's focus on a brief mindfulness-based self-compassion intervention stands out as a resource-efficient and practical approach to addressing aggression in adolescents. This concise intervention's potential effectiveness offers the promise of a more accessible and cost-effective approach to addressing adolescent aggression, which is critical in our resource-constrained world. The study determined that the brief intervention is efficacious, enabling its adaptation and implementation in educational institutions, juvenile justice programs, and community organizations that work with belligerent adolescents. Due to its versatility, the conclusions of the study can be directly applied to real-world issues. The salient feature of this method is in its explicit targeting of adolescent aggression. By prioritizing self-compassion and mindfulness, this program aids in the regulation of emotions and reduces aggression among young individuals. Effective interventions have the potential to improve the psychological well-being, emotional control, and interpersonal connections of adolescents who display aggressive behavior. This study has the potential to make mindfulness-based self-compassion practices more easily available to a greater number of adolescents. This might lead to the development of practical and cost-effective solutions that promote emotional well-being and decrease aggressiveness. These strategies would have long-lasting advantages.

ELIGIBILITY:
Inclusion Criteria:

1. Students' age range of 13 to 19 years
2. symptoms of aggression.

Exclusion Criteria:

Students who are not willing to participate

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Psychological Wellbeing | 1 Month
  after the intervention (mindfullness) students shows the significant improvement in their psychological wellbeing

CONTACTS AND LOCATIONS:
Locations (1):
- Muhammad Rizwan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The ethical committee of FJWU Rawalpindi approved the research topic in the first phase. The principals of the government and private schools in Rawalpindi granted permission for the data collection. Prior to the commencement of the study, we debriefed the participants about the research topic and its conduct modalities. Participants were approached by purposive sampling. We obtained informal consent from both the students and the parents.
  3.7.2 Phase II In the second phase of the research, the participants were randomly assigned to the control and intervention groups by using software. The interventional group exposed participants to Urdu-adapted and translated mindfulness-based self-compassion training. However, the control group either maintained their usual routine or standard care, or received a non-specific intervention. After the successful completion of mindfulness-based self-compassion training, both groups were evaluated. Pre- and post-assessment results were assessed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six Month